CLINICAL TRIAL: NCT03815929
Title: Impact of Individualized Estrogen Therapy on Cardiovascular Disease Risk Parameters in Young Women After Bilateral Oophorectomy: A Randomized Controlled Trial
Brief Title: Oophorectomy, Estrogen Therapy and Cardiovascular Disease Risk in Young Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ekta Kapoor, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-007999
Record Dates: First submitted 2019-01-17; First posted 2019-01-24 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Risk Reduction
Keywords: Hormone therapy; Pre-menopausal Oophorectomy; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Ortho Evra

STUDY DESIGN:
Intervention Model Description: Subject be placed into three different study arms. Subjects undergoing surgery will be randomized to receive either standard hormone therapy or individualized hormone therapy. These arms will be compared against each other as well as a third arm of healthy timed-control subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Standard replacement therapy regimen (Active Comparator): 100 mcg transdermal estradiol patch (or equivalent oral dose)
  Interventions: Drug: Estradiol 100 Micrograms Patch
- Titrated replacement therapy regimen (Active Comparator): Transdermal estradiol patch (or equivalent oral dose) titrated to achieve pre-menopausal estradiol level
  Interventions: Drug: Estradiol Patch
- Timed Control Group (No Intervention): Healthy age-matched subjects not on hormone therapy

INTERVENTIONS:
Drug: Estradiol 100 Micrograms Patch — Standard
  Arms: Standard replacement therapy regimen
Drug: Estradiol Patch — Individualized
  Arms: Titrated replacement therapy regimen

SUMMARY:
Researchers are trying to assess the appropriate dose of estrogen for decreasing the risk of cardiovascular disease in women who have removal of their ovaries at a young age, before the age of 46 years.

DETAILED DESCRIPTION:
Baseline Study Visit: Subjects will report for the Baseline Study Day in an 8 hour fasting state (water only) and refrain from heavy exercise, caffeine, and alcohol for 24 hours. The participant will undergo study specific procedures including a urine pregnancy test if they are of child bearing potential. Participants will also complete a set of questionnaires. After the completion of the study tests, participants will be offered a meal.

Participants scheduled for surgery to remove their ovaries: after the surgery subjects will be randomized to one of two groups. They will receive the standard dose of the hormone (estrogen) patch, generally prescribed to patients after removal both ovaries. Or sent home on the standard dose hormone patch, hormone levels will be tested every 3-4 weeks, and patch dose adjusted until the estrogen level is reached that results in the hormone levels of a young woman before menopause. In order to check hormones, subjects will be able to choose to have a lab kit sent to them and have the draw done locally, or can come in person.

Participants will also receive a second hormone prescription if they have an intact uterus to protect the lining of the uterus from the effects of using estrogen alone.

6-Month Study Visit: Subjects will be asked to come back and repeat most of the study specific tests from the baseline study visit that will take about 5 hours.

1-Year Study Visit: Subjects will be asked to come back for the final visit and will repeat all the study tests done at baseline visit. This visit will take about 5 hours.

Control Group: Healthy subjects serving as controls to see how measures change over time will not undergo a surgery or be given estrogen. These healthy subjects will return after the baseline visit to repeat study visits at 6 and 12-months.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women undergoing (or completion of a) bilateral oophorectomy for non-malignant diagnoses at Mayo Clinic, Rochester; or premenopausal women not undergoing the procedure for the timed control group
* Currently between the ages of 21- 45 years
* Able to participate fully in all aspects of the study
* Able to understand and sign the informed consent.

Exclusion Criteria:

* History of hepatic, renal, or hematological diseases
* History of venous thromboembolism; peripheral vascular disease; coronary artery disease; stroke/neurovascular disease
* Chemotherapy or radiation therapy in the preceding 3 months
* Current tobacco use
* Current use of medication that alters autonomic or vascular function (e.g. tricyclic antidepressants, α-blockers, β-blockers, etc.) or aromatase inhibitor/tamoxifen therapy
* Contra-indication to estrogen use
* Current or previous diagnosis of breast and endometrial cancer
* For Timed Controls: Are currently pregnant or lactating, or are of child-bearing potential or are likely to become pregnant during the study and unwilling to use contraception; Acceptable forms include:Barrier methods (such as a condom or diaphragm) used with a spermicide (a foam, cream, or gel that kills sperm), Copper Intra Uterine Device, Hysterectomy, Tubal ligation, Abstinence (no sex)
* Any condition or factor judged by the investigator to preclude participation in the study

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ekta Kapoor, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20451789

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Replacement Therapy Regimen | Titrated Replacement Therapy Regimen | Timed Control Group
Started | 15 | 15 | 5
Baseline | 15 | 15 | 5
6-month | 12 | 12 | 4
12-month | 11 | 12 | 4
Completed | 11 | 12 | 4
Not Completed | 4 | 3 | 1
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Physician Decision | 2 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Replacement Therapy Regimen | Titrated Replacement Therapy Regimen | Timed Control Group | Total
Number analyzed (Participants) | 15 | 15 | 5 | 35
Age, Customized [Count of Participants; unit: Participants]
  21-45 years old | 15 | 15 | 5 | 35
  >46 years old | 0 | 0 | 0 | 0
  < 20 years old | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 5 | 35
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 5 | 35

OUTCOME MEASURES:

1. Primary Outcome: Arterial Stiffness
Description: Augmented pressure, a measure of arterial stiffness was recorded through high-fidelity pressure waveforms and compared at planned time frames
Time Frame: Baseline, 6 months, and 12 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Standard Replacement Therapy Regimen | Titrated Replacement Therapy Regimen | Timed Control Group
Number analyzed (Participants) | 10 | 12 | 4
mm Hg
  Baseline augmented pressure | 10.1 (6.9) | 14.8 (4.3) | 6.4 (3.7)
  6 months augmented pressure | 12.7 (6.0) | 16.8 (6.4) | 5.1 (3.1)
  12 months augmented pressure | 12.9 (6.7) | 17.3 (7.2) | 6.5 (4.0)

2. Secondary Outcome: Mean Blood Pressure Reactivity to Isometric Hand Grip Exercise
Description: Change in mean blood pressure in response to isometric hand grip exercise (30% maximum voluntary contraction)
Time Frame: Baseline, 6 months, and 12 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Standard Replacement Therapy Regimen | Titrated Replacement Therapy Regimen | Timed Control Group
Number analyzed (Participants) | 9 | 11 | 4
mm Hg
  baseline mean blood pressure reactivity | 11.6 (4.6) | 11.4 (5.9) | 8.3 (3.5)
  6-month mean blood pressure reactivity | 11.7 (5.0) | 15.3 (5.3) | 10.7 (2.6)
  12-month mean blood pressure reactivity | 16.2 (7.1) | 12.4 (7.6) | 13.9 (9.9)

3. Secondary Outcome: Mean Blood Pressure Reactivity to Cold Stress
Description: Maximum change in mean blood pressure during 3-minute cold pressor test (immersing hand up to wrist in ice water while changes in blood pressure monitored)
Time Frame: Baseline, 6 months, and 12 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Standard Replacement Therapy Regimen | Titrated Replacement Therapy Regimen | Timed Control Group
Number analyzed (Participants) | 8 | 10 | 4
mm Hg
  Baseline mean blood pressure reactivity | 22 (10) | 20 (9) | 20 (8)
  6-month mean blood pressure reactivity | 21 (13) | 25 (9) | 18 (5)
  12-month mean blood pressure reactivity | 26 (12) | 25 (7) | 17 (3)

4. Secondary Outcome: Changes in Whole Body Fat
Description: Measurements of whole-body fat using Dual energy x-ray absorptiometry (DXA)
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: gm
Arm/Group | Standard Replacement Therapy Regimen | Titrated Replacement Therapy Regimen | Timed Control Group
Number analyzed (Participants) | 10 | 15 | 4
gm
  Baseline total body fat | 30712 (12958) | 43363 (26212) | 199936 (14221)
  12-month total body fat | 31868 (18020) | 42660 (25938) | 16735 (3114)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Standard Replacement Therapy Regimen | Titrated Replacement Therapy Regimen | Timed Control Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/15 | 2/15 | 0/5
Other Adverse Events (participants affected / at risk) | 3/15 | 11/15 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Replacement Therapy Regimen (N=15) | Titrated Replacement Therapy Regimen (N=15) | Timed Control Group (N=5)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia of unknown etiology after planned oophorectomy & liver procedure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Liver Infarct (extended hospital stay) (General disorders) | 0 (0) | 1 (1) | 0 (0)
non-focal Bile leak from disease resection (extended hospital stay) (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Replacement Therapy Regimen (N=15) | Titrated Replacement Therapy Regimen (N=15) | Timed Control Group (N=5)
Rash at patch site (General disorders) | 1 (1) | 1 (1) | 0 (0)
Passed out after blood draw at CRTU (General disorders) | 0 (0) | 1 (1) | 0 (0)
Moderate bilateral pleural effusion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian Cancer Stage IIIc high grade Serious Carcinoma (General disorders) | 0 (0) | 1 (1) | 0 (0)
COVID 19 (General disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased Libido (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder Issues (General disorders) | 0 (0) | 1 (1) | 0 (0)
Headache/vomitting/allergic reaction to MRI (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal cuff dehiscence (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pain with intercourse, vaginal dryness, and low sex drive (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine with vomitting during blood pressure regulation baseline testing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Itching from patch site (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal cuff dehiscence with infection (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Estradiol gives burnt taste in mouth (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT03815929/Prot_SAP_000.pdf